CLINICAL TRIAL: NCT02255526
Title: BodyGuardian Respiration and Activity Validation Testing
Status: Completed | Type: Observational
Sponsor: Preventice (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 14-004034
Record Dates: First submitted 2014-09-26; First posted 2014-10-02 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Healthy volunteers between the ages of 18 and 80 will wear BodyGuardian remote monitoring system to help validate respiration and activity levels.
  Interventions: Device: BodyGuardian
- Heart Failure: Heart failure patients between the ages of 18 and 80 will wear BodyGuardian remote monitoring system to help validate respiration and activity levels.
  Interventions: Device: BodyGuardian

INTERVENTIONS:
Device: BodyGuardian — BodyGuardian (BG) device will be worn by all subjects to determine accuracy of respiration and activity levels monitored by BG

SUMMARY:
This project will compare BodyGuardian (BG) device measurements of breathing and activity levels to the gold standard measurement techniques of gas exchange using a mouthpiece connected to flow and gas analyzers measures for breathing and metabolic rate (indirect calorimetry) for activity, We are hopeful these comparisons will help us improve upon the measurements being made in the current version of the BG device.

DETAILED DESCRIPTION:
BodyGuardian remote monitoring system is an FDA 510 cleared device used to perform remote monitoring of cardiac patients. BodyGuardian (BG) is a novel remote care platform. It incorporates an adhesive strip sensor with in-built electrodes attached to a rechargeable module that can determine an ECG signal and bio impedance. The module also has a 3-way accelerometer. ECG, physical activity and respiration can be assessed using these sensors. Although ECG data is reliable, there are doubts regarding the clinical meaning and validity of the activity and respiration data.

The BG reports respiration rate and activity level (on a scale of 0 to 100). This data is being used as input into other clinical algorithms including onboard ECG arrhythmia detection as well as clinical care algorithms for heart failure decompensation prediction.

Respiration data is not uniformly reported and there is still doubt regarding its validity. BG breathing measurements will be compared to gold standard measurement techniques of gas exchange using a mouthpiece connected to flow and gas analyzer. Activity data is reported but the investigators do not know how the value translates into clinically used objective parameters of activity e.g. METS. BG activity measurements will be compared to the gold standard activity measurements using metabolic rate (indirect calorimetry)

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers between the ages of 18-80
* Heart Failure Patients/ Volunteers between the ages of 18-80

Exclusion Criteria:

* Healthy - Non Ambulatory. With Pacemaker. Not able to sign consent.
* Hospitalized in last 6 months for fractures, myocardial infarcts, cancer related surgery, chemo therapy. Allergies to silicone or acrylic hydrogel adhesives, fragile skin, and/or pregnancy
* Heart Failure - Non Ambulatory. With Pacemaker. Not able to sign consent.
* Hospitalized in last 6 months for fractures, cancer related surgery, chemo therapy.
* Allergies to silicone or acrylic hydrogel adhesives, fragile skin, and/or pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers and Heart Failure patients
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of successful breathing and activity measurements recorded by BG | 1 year
  Measurements of BG breathing (rate and patterns) with impedance and accelerometry compared to gold standards using a mouthpiece connected to flow and gas exchange analyzers.
  BG activity level measurements based on accelerometry compared to gold standard measures of metabolic rate (indirect calorimetry).

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Johnson, Ph.D., Principal Investigator — Mayo Clinic, Rochester, MN
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Not an applicable study under section 801